CLINICAL TRIAL: NCT07250828
Title: Therapeutic Efficacy and Feasibility Study of Abbott's BurstDR Spinal Cord Stimulators Technology for Painful Diabetic Neuropathy (PDN)
Brief Title: Efficacy and Feasibility of BurstDR SCS in Painful Diabetic Neuropathy
Acronym: ABBT DPN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TriCity Research Center (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS-25-ABT-002; ABT-002 (Other: TriCity Research Center)
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Painful Diabetic Neuropathy (PDN); Diabetic Neuropathy; Neuropathic Pain; Chronic Pain
Keywords: Painful Diabetic Neuropathy; Diabetic Neuropathy; Neuropathic Pain; Spinal Cord Stimulation; BurstDR; Proclaim XR; Eterna SCS; Neuromodulation
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm study in which all participants receive BurstDR spinal cord stimulation using Abbott Proclaim XR or Eterna systems.
Masking Description: Open-label study. No parties are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test Group [Burst DR SCS] (Experimental): Participants receive BurstDR spinal cord stimulation delivered through Abbott Proclaim XR or Eterna systems, beginning with a temporary trial followed by permanent implantation for responders.
  Interventions: Device: BurstDR Spinal Cord Stimulation

INTERVENTIONS:
Device: BurstDR Spinal Cord Stimulation — Participants receive BurstDR spinal cord stimulation delivered through Abbott Proclaim XR or Eterna spinal cord stimulator systems in a standard of care routine. The intervention includes a one-week temporary SCS trial using percutaneous leads, followed by permanent implantation of the Proclaim XR or Eterna implantable pulse generator for participants who experience meaningful pain relief during the trial. Device programming and follow-up assessments follow standard clinical practice.
  Other Names: Proclaim; Eterna; Burst DR; Spinal Cord Stimulator

SUMMARY:
This prospective, single-arm clinical study evaluates the therapeutic efficacy and feasibility of BurstDR spinal cord stimulation (SCS) using Abbott's Proclaim XR and Eterna systems in patients with painful diabetic neuropathy (PDN). Adults with confirmed PDN will undergo a one-week temporary SCS trial, and those achieving meaningful improvement (≥50% reduction in average pain on the Visual Analog Scale) will proceed to permanent implantation. Outcomes will be assessed at baseline, end of trial, and at 1-, 3-, and 6-month follow-up visits using validated instruments including VAS, DN4, DQoL, PSQ-3, the Patient Global Impression of Change, and the Clinician Global Impression of Change. All procedures follow standard clinical practice for SCS therapy. The study aims to characterize real-world effectiveness, patient-reported outcomes, feasibility of implementation, and device-related safety in a rural PDN population.

DETAILED DESCRIPTION:
This investigator-initiated, post-market clinical study is designed to evaluate the efficacy, feasibility, and safety of BurstDR spinal cord stimulation (SCS) for the management of painful diabetic neuropathy (PDN) using Abbott's Proclaim XR and Eterna implantable pulse generator systems. The SCS systems used in this study are FDA-approved for PDN, and all clinical procedures-including the percutaneous trial phase and permanent implantation-are performed according to standard-of-care practice by experienced clinicians.

Eligible participants are adults aged 19 years or older with confirmed diabetic neuropathy (via EMG or skin biopsy), neuropathic pain severity meeting VAS ≥6 and DN4 ≥4, failure of conventional medical therapy, and suitability for SCS treatment. After informed consent, participants will complete baseline assessments followed by a temporary one-week SCS trial with BurstDR stimulation. Participants who experience meaningful pain reduction during the trial will proceed to permanent implantation. Follow-up assessments occur at 1, 3, and 6 months after implantation, during which validated patient-reported outcomes and clinician-reported measures will be collected. Adverse events, device-related complications, therapy discontinuations, and protocol deviations will be monitored and documented.

The study's primary objective is to determine the proportion of participants achieving ≥50% pain reduction on the Visual Analog Scale at follow-up visits. Secondary objectives evaluate changes in diabetes-related quality of life (DQoL), neuropathic symptoms (DN4), sleep interference (PSQ-3), and patient and clinician impression of change. Tertiary objectives assess feasibility parameters including recruitment rates, retention, protocol adherence, and safety outcomes. Data will be captured and stored using a HIPAA-compliant, 21 CFR Part 11-validated Clinical Trial Management System. The study is conducted at TriCity Research Center with IRB oversight and is funded by Abbott, which has no role in study design, data analysis, or publication decisions.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older.
* Diagnosis of diabetic peripheral neuropathy (DPN) confirmed by nerve conduction study (EMG/NCS) or skin biopsy.
* Persistent neuropathic pain in the lower extremities for ≥6 months.
* Average baseline pain score of ≥6 on the Visual Analog Scale (VAS).
* DN4 score ≥4, indicating neuropathic pain characteristics.
* Inadequate pain relief with conventional medical therapy, including at least two classes of analgesic or neuropathic pain medications (e.g., gabapentinoids, SNRIs, TCAs, opioids).
* Candidate for spinal cord stimulation based on clinical evaluation by the treating physician.
* Able and willing to comply with all trial procedures and follow-up visits.
* Able to provide written informed consent in English or in an IRB-approved translated language.

Exclusion Criteria:

* Prior spinal cord stimulator implantation or previous SCS trial that was unsuccessful.
* Contraindications to SCS placement, including:
* Active systemic infection or local infection at planned needle entry site
* Bleeding disorders or inability to temporarily discontinue anticoagulation if required
* Known allergy to device materials or components
* Severe uncontrolled medical conditions that increase surgical risk, including:
* Unstable cardiovascular disease
* Severe renal or hepatic dysfunction
* Uncontrolled diabetes (e.g., HbA1c > 10%)
* Severe or uncontrolled psychiatric illness that, in the investigator's judgment, may interfere with study compliance.
* Current substance use disorder, including active opioid misuse or illicit drug use, based on clinician assessment.
* Pregnancy or planning to become pregnant during the study period.
* Life expectancy less than 12 months.
* Participation in another interventional clinical trial that may confound results or interfere with study procedures.
* Any condition that, in the investigator's opinion, makes the participant unsuitable for SCS therapy or the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
VAS Change Baseline to 6 Month | 1 month, 3 months, and 6 months
  Pain will be assessed using the Visual Analog Scale (VAS). The primary endpoint is the proportion of participants who achieve at least a 50% reduction in average VAS pain score from baseline to each follow-up visit after permanent implantation.

SECONDARY OUTCOMES:
Diabetes QoL Change Baseline to 6 Months | 1 month, 3 months, and 6 months after permanent implantation
  Quality of life will be assessed using the Diabetes Quality of Life (DQoL) questionnaire. The outcome is the change in total DQoL score from baseline to each follow-up visit. Clinically meaningful improvement is defined as a ≥0.05-point increase in the DQoL index.
Change in DN4 neuropathic pain score | 1 month, 3 months, and 6 months after permanent implantation
  Neuropathic symptoms will be measured using the DN4 questionnaire. The outcome is the change in DN4 score from baseline to follow-up. Clinically meaningful improvement is defined as a ≥2-point reduction in DN4 score.
Change in pain-related sleep interference (PSQ-3) | 1 month, 3 months, and 6 months after permanent implantation
  Sleep interference will be assessed using the Pain and Sleep Questionnaire-3 item (PSQ-3). The outcome is the percentage reduction in PSQ-3 score from baseline to follow-up. Clinically meaningful improvement is defined as a ≥30% reduction.

CONTACTS AND LOCATIONS:
Locations (1):
- Grand Island Pain Relief Center, Grand Island, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided